CLINICAL TRIAL: NCT05020860
Title: A Phase II Trial to Correlate Early Clinical Response to Pathologic Outcome With Neoadjuvant Systemic Therapy in Patients With Early Stage Breast Cancer
Brief Title: Correlation of Clinical Response to Pathologic Response in Patients With Early Breast Cancer
Acronym: RESPONSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Professor, Baylor Breast Care Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-50349
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Neoplasm; Breast Cancer Female; Breast Cancer Invasive; Breast Cancer Stage II; Breast Cancer Stage III; Triple Negative Breast Cancer; Hormone Receptor-positive Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Neoplasms; Estrogen Receptor-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Trastuzumab; pertuzumab; Doxorubicin; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Triple Negative Breast Cancer (for tumors > 5 cm) (Active Comparator): Paclitaxel IV plus carboplatin IV (+/- pembrolizumab IV) (4 cycles total), followed by doxorubicin IV plus cyclophosphamide IV (+/- pembrolizumab IV) (4 cycles total)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Pembrolizumab
- Triple Negative Breast Cancer (for tumors < 5 cm) (Active Comparator): Paclitaxel IV (4 cycles total), followed by doxorubicin IV plus cyclophosphamide IV (4 cycles total)
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- HER2-Positive Breast Cancer (Active Comparator): Paclitaxel IV plus Trastuzumab IV plus Pertuzumab IV (or PHESGO) (4 cycles total), followed by doxorubicin IV plus cyclophosphamide IV administered (4 cycles total)
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Pertuzumab/Trastuzumab/Hyaluronidase-zzxf
- Hormone Receptor Positive Breast Cancer (Active Comparator): Paclitaxel IV plus Carboplatin IV (4 cycles total), followed by doxorubicin IV plus cyclophosphamide IV (4 cycles total)
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 IV administered on Days 1, 8, 15 of each 21-day cycle
  Other Names: Taxol
Drug: Carboplatin — Carboplatin AUC 1.5 IV administered on Days 1, 8, 15 of each 21-day cycle
  Arms: Triple Negative Breast Cancer (for tumors > 5 cm)
Drug: Trastuzumab — Trastuzumab 8 mg/kg loading dose, followed by 6 mg/kg maintenance dose, administered on Day 1 of each 21-day cycle
  Other Names: Herceptin
  Arms: HER2-Positive Breast Cancer
Drug: Pertuzumab — Pertuzumab 840 mg loading dose, followed by 420 mg maintenance dose, administered on Day 1 of each 21-day cycle
  Other Names: Perjeta
  Arms: HER2-Positive Breast Cancer
Drug: Doxorubicin — 60 mg/m2 IV administered on Day 1 of each 14-day cycle
  Other Names: Adriamycin
Drug: Cyclophosphamide — 600 mg/m2 IV administered on Day 1 of each 14-day cycle
  Other Names: Cytoxan
Drug: Pembrolizumab — Either 200 mg IV administered on Day 1 of Cycles 1-4, or 400 mg IV administered on Day 1 of Cycles 1 and 3 of the paclitaxel/carboplatin regimen.
  400 mg on Day 1 of Cycles 1 and 4 of the dose-dense AC regimen.
  Other Names: Keytruda
  Arms: Triple Negative Breast Cancer (for tumors > 5 cm)
Drug: Pertuzumab/Trastuzumab/Hyaluronidase-zzxf — Can be used in place of separate IV formulations of pertuzumab and trastuzumab. 1200 mg pertuzumab/600 mg trastuzumab/30,000 U hyaluronidase administered subcutaneously on Day 1 of the first cycle, followed by a maintenance dose of 600 mg pertuzumab/600 mg trastuzumab/20,000 U hyaluronidase administered subcutaneously every 3 weeks.
  Other Names: PHESGO
  Arms: HER2-Positive Breast Cancer

SUMMARY:
The purpose of this study is to learn whether clinical response (the amount a tumor shrinks based on imaging or tumor measurements obtained by physical exam) predicts pathologic response (the amount of tumor remaining when surgery is performed) in participants with breast cancer who are receiving chemotherapy prior to surgery.

DETAILED DESCRIPTION:
Neoadjuvant therapy was first introduced to improve surgical outcomes of breast cancer and to be able to assess the pathological responsiveness to therapy at the time of surgery. Over time, it became a useful experimental platform in clinical research in breast cancer, and in recent years became an important part of standard management of certain subtypes and clinical stages in breast cancer.

It has been long established that patients who achieve pathologic complete response (pCR, i.e., the absence of any cancer in the tissue removed during surgery) after receiving neoadjuvant treatment have better outcomes than those who don't, especially in HER2+, and triple-negative breast cancer (TNBC). Many reports add aggressive ER+ breast cancer to these groups. So far, the only way to know whether a patient achieved pCR is to give them a full course of therapy and then proceed to surgery.

One of the areas that has attracted significant research interest has been the effort to develop early predictors of pCR. This way, treatment can be tailored in the future to each patient and each tumor and can spare patients ineffective therapy. Some of these predictors include tissue biomarkers, blood based biomarkers, and imaging biomarkers.

It has been observed in neoadjuvant clinical trials that many patients have an impressive early clinical response to treatment after 1-2 cycles of treatment. Anecdotally, many of those patients go on to have a pCR at the time of surgery. This observation, if validated in a prospective clinical trial, may lead to a simple, inexpensive way to assess tumor responsiveness and predict pCR using clinical exam and simple imaging.

Using imaging or molecular changes to predict pCR will also be explored in this study. A consortium of investigators will be studying image analysis and proteogenomic changes early in the course of treatment to predict clinical response specifically in participants with TNBC. Only participants with TNBC will be required to undergo a research biopsy and research MRI prior to starting treatment, and again after the first cycle of treatment.

The investigators therefore hypothesize that absence of early clinical response, defined as at least a 30% reduction in the size of the breast tumor by Day 21 of treatment (as measured by either imaging or clinical exam), will be associated with absence of pCR at the time of surgery, in 3 subtypes of breast cancer - TNBC, HER2+, high-risk ER+.

All treatment in this study is standard of care (non-investigational).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, and legally able to provide informed consent. Both men and women are eligible.
* Histologically confirmed, invasive breast cancer. Tumor may be triple negative (as defined by ASCO-CAP guidelines), HER2-positive (as defined by ASCO-CAP guidelines), or high-risk estrogen receptor positive (as defined by ASCO-CAP guidelines).

To be considered "high risk," at least 2 of the following criteria must be met: 1) histologic grade 3; 2) patient age 50 or less; 3) ER Allred score < 6; 4) Ki-67 ≥ 30%.

* Tumors must be at least 2 cm by clinical exam or ultrasound
* Bilateral breast cancers are allowed if the following criteria are met: 1) A lesion on one side (meeting the criteria above) is designated as the index lesion on which study assessments will be performed, and 2) the same treatment regimen is appropriate for both cancers as determined by the treating physician.
* ECOG performance status of 0 or 1
* Left ventricular ejection fraction (LVEF) ≥ the institutional lower limit of normal, as assessed by echocardiogram or Multigated Acquisition (MUGA )scan.
* Adequate organ function, as determined by the following parameters:

  * Absolute Neutrophil Count (ANC) ≥ 1200/mm3
  * Platelets ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ institutional upper limit of normal (ULN), unless patient has Gilbert's disease or similar syndrome
  * Alkaline phosphatase (ALP) ≤ 2.5 x institutional ULN
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 1.5 x institutional ULN
  * Serum creatinine ≤ institutional ULN
* The participant, if of childbearing potential, is willing to use effective, non-hormonal contraception while on treatment.
* Participation in a concurrent clinical trial is permitted, with Principal Investigator approval.

Exclusion Criteria:

* Definitive clinical or radiologic evidence of Stage IV disease
* Inflammatory breast cancer
* Participants who are pregnant or lactating
* History of an excisional biopsy or lumpectomy performed prior to study entry
* Prior treatment with anthracyclines for any malignancy.
* Prior treatment for currently diagnosed breast cancer (i.e., endocrine therapy, chemotherapy, targeted therapy, or radiation.
* History of cardiac disease that would preclude the use of drugs included in these treatment regimens. This includes, but is not limited to:

  * Angina pectoris requiring the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with documented compromise in cardiac function
  * Symptomatic pericarditis
  * Documented cardiomyopathy
  * History of documented congestive heart failure (CHF)
  * Myocardial infarction documented by elevated cardiac enzymes, or persistent regional wall abnormalities on assessment of left ventricular function.
* Current HIV, hepatitis B, or hepatitis C infection
* History of non-breast malignancies (with the exception of in situ cancers treated only by local excision, and basal cell or squamous cell carcinoma of the skin) within 5 years prior to enrollment.
* Any other non-malignant systemic disease that would preclude treatment with any of the treatment regimens or prevent required follow-up.
* Any psychiatric or addictive disorders, adverse social situations, or other medical conditions that, in the opinion of the investigator, would preclude the patient from meeting study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Tumor Measurement vs. Pathologic Response | Baseline and at surgery (after 20 weeks)
  Clinical tumor measurements are tumor measurements obtain via imaging (mammogram or ultrasound) or by physical exam. Pathologic response is the amount of tumor remaining at the time of surgery, as determined by the pathologist.

SECONDARY OUTCOMES:
Pathologic Complete Response Rate in each Breast Cancer Subtype | 20 weeks
  A pathologic complete response (pCR) means that there is no residual invasive cancer identified in the tissue removed at surgery. The frequency of pCR will be estimated for each breast cancer subtype (triple negative, hormone receptor positive, and HER2-positive)
Predictive value of clinical response following 1 cycle of chemotherapy to predict pathologic complete response | 20 weeks
  This aims to determine whether a 30 percent reduction in tumor size (as measured by physical exam or imaging) following one cycle of chemotherapy can predict whether a patient will have no residual invasive cancer at the time of surgery

OTHER OUTCOMES:
Change in circulating tumor DNA (ctDNA) levels from baseline to surgery | 20 weeks
  ctDNA is DNA from a tumor circulating in a patient's bloodstream. The goal of this is to determine whether a decrease in ctDNA levels (as measured from baseline to surgery) correlates to clinical and/or pathologic response

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Harris Health System - Smith Clinic, Houston, Texas
  - O'Quinn Medical Tower - McNair Campus - Dan L Duncan Comprehensive Cancer Center, Houston, Texas